CLINICAL TRIAL: NCT00300742
Title: Topiramate for the Treatment of Alcohol Dependent Binge-Eating Disordered Individual
Brief Title: Topiramate for the Treatment of Alcohol Dependent Binge-Eating Disordered Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Addiction Research and Education, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12069
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2012-02

CONDITIONS: Alcohol Dependence; Binge Eating
Keywords: drinking; eating; obesity; alcohol; binge eating
MeSH Terms: conditions — Alcoholism; Bulimia; Obesity | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topiramate (Experimental): Drug: Topiramate Other Name for Topiramate: Topamax
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate up to 300 mg per day.
  Other Names: Topamax

SUMMARY:
The purpose of this study is to test the feasibility of using topiramate to reduce binge eating and drinking episodes in alcohol dependent individuals with comorbid binge eating disorder.

DETAILED DESCRIPTION:
Research has shown an alarming coincidence of binge eaters also reporting serious alcohol abuse. Evidence has shown this population to have higher rates of psychiatric comorbidity, higher caloric intakes during meals, higher rates of tobacco use, more frequent binge episodes, and an earlier age of onset for binge eating and alcohol abuse. It is believed that topiramate may reduce binge eating and has been found helpful in reducing the cravings associated with alcohol consumption.

This study is to test the feasibility of administering topiramate to individuals with alcohol dependence and binge eating disorder. This will involve determining the adequacy of the amount of assessment and scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Males and females that have given written informed consent.
* Good physical health as confirmed by a complete physical examination, vital signs including an EKG within normal limits, laboratory screening tests within acceptable parameters (see exclusion criteria), as well as a baseline psychiatric history
* Diagnosis of alcohol dependence and binge eating disorder.
* Subjects must have 3 or more binge days per week in the 2-week period prior to Screen.
* Subjects may have uncomplicated and well-controlled Type II diabetes and/or hypertension that has been well controlled by diet and/or oral agent therapy for at least 3 months prior to screen.
* Provide evidence of stable residence in the last month.
* The pregnancy test for females at intake must be negative. The female patients must either be sterile, post menopausal, or practicing an acceptable form of contraception.
* Literate in English and able to read, understand, and complete the ratings scales and questionnaires accurately, follow instructions, and make use of the behavioral treatment.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Any current DSM-IV psychiatric diagnosis other than alcohol, nicotine dependence or binge eating disorder
* Subjects who have begun to receive formal psychotherapy (cognitive-behavioral therapy, interpersonal therapy, dietary behavioral therapy*, or self-guided cognitive-behavioral) for binge-eating disorder or any other psychiatric disorder within 30 days prior to Screen. Subjects who have been engaged in formal psychotherapy for a longer period of time and plan to maintain therapy will be judged on a case-by-case basis.

  * Formal dietary behavioral therapy applies to therapy where the subject is diagnosed with an eating disorder and/or the health case provider is billing for costs of therapy (will be considered on a case-by-case basis if started within 30 days of Screen. Subjects engaged in dietary for obesity only (e.g., Jenny Craig, Weight Watchers, Overeater's Anonymous) should discontinue therapy prior to study entry (no washout applies).
* Clinically significant laboratory screening test.
* Clinically significant cardiovascular disease on a 12 lead EKG.
* Symptomatic coronary artery disease or peripheral vascular disease.
* Malignancy or history of malignancy within the past 5 years (except basal cell carcinoma).
* Clinically significant neurological disease.
* Clinically significant renal disease or impaired renal function as defined by subjects with an estimated creatinine clearance of less than 60 mL/min.
* Severe withdrawal symptoms which in the physicians' opinion requires inpatient treatment or severe or life-threatening adverse reactions to medications either in the past or during this clinical trial.
* Female patients who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study.
* Members of the same household.
* History of severe hypersensitivity to any medication or environmental allergens.
* Subjects with prior non-response to topiramate for the treatment of binge-eating and or alcohol disorder following an adequate trial of this medication
* Subjects who have been previously treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud, MD, Principal Investigator — University of Virginia, Department of Psychiatric Medicine
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Charlottesville and Richmond between September 2006 to February 2007.
Groups:
- Topiramate/BBCET: Escalating dose of up to 300 mg/day of Topiramate
Period: Overall Study
Arm/Group | Topiramate/BBCET
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10.46422)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Study Requirements: Attendance at Treatment Sessions
Time Frame: up to 12 weeks
Measure: Number; unit: participants
Groups:
- Topiramate/BBCET: Patients receiving an escalating dose of up to 300 mg/day of Topiramate, plus BBCET (Brief Behavioral Compliance Enhancement Treatment)
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
participants
  Number of subjects completed through Visit 4 | 5
  Number of subjects completed through Visit 12 | 3

2. Primary Outcome: Mean Drinks Per Day at Baseline vs. Visit 12
Description: Mean drinks per day at baseline vs. Visit 12 measured by self report on timeline follow-back (TLFB) calendars in conjunction with the subject's daily diary
Time Frame: up to 24 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Drinks/day
Groups:
- Topiramate/BBCET: Escalating dose of up to 300 mg/day of Topiramate, plus BBCET (Brief Behavioral Compliance Enhancement Treatment)at 12 weekly visits following the initial baseline and randomization visits
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
Drinks/day
  Mean drinks per day at baseline | 10.95 (13.85)
  Mean drinks per day at Visit 12 | 0.68 (1.13)

3. Primary Outcome: Mean Percent Days Abstinent Per Week at Baseline vs. Visit 12
Description: Mean percent days abstinent per week at baseline vs. Visit 12 measured by self report on timeline follow-back (TLFB) calendars in conjunction with the subject's daily diary
Time Frame: up to 24 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Mean percent days abstinent per week
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
Mean percent days abstinent per week
  Mean percent days abstinent per week at baseline | 20 (21.67)
  Mean percent days abstinent per week at Visit 12 | 76.2 (7.14)

4. Primary Outcome: Mean Binge Eating Episodes Per Week at Baseline vs. Visit 12
Description: Mean binge eating episodes per week at baseline vs. Visit 12 measured by self report on timeline follow-back (TLFB) calendars in conjunction with the subject's daily diary
Time Frame: up to 24 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Binge eating episodes/week
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
Binge eating episodes/week
  Mean weekly binge eating episodes at baseline | 3.7 (2.11)
  Mean weekly binge eating episodes at Visit 12 | 1 (1.7)

5. Primary Outcome: Compliance With Study Requirements: Topiramate Level
Description: Number of subjects who escalated to the maximum dose of 300 mg of topiramate/day
Time Frame: up to 12 weeks
Population: This is the number of participants who reached the dose of 300 mg of topiramate
Measure: Number; unit: participants
Arm/Group | Topiramate/BBCET
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Arm/Group | Topiramate/BBCET
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No